CLINICAL TRIAL: NCT03994666
Title: Cell Therapy in Critical Limb Ischemia by Implantation of Allogeneic Umbilical Cord-derived Mesenchymal Stem Cells
Brief Title: Cell Therapy in Critical Limb Ischemia
Acronym: CLI
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PO19059
Record Dates: First submitted 2019-06-04; First posted 2019-06-21 (Actual); Last update posted 2019-06-21 (Actual); Status verified 2019-06

CONDITIONS: Critical Limb Ischemia
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- simple dose (Experimental)
  Interventions: Biological: allogeneic umbilical cord-derived mesenchymal stem cells
- double dose (Experimental)
  Interventions: Biological: allogeneic umbilical cord-derived mesenchymal stem cells
- placebo (Placebo Comparator)
  Interventions: Biological: Placebo (NaCl)

INTERVENTIONS:
Biological: allogeneic umbilical cord-derived mesenchymal stem cells — Injection of mesenchymal stem cells
  Arms: double dose; simple dose
Biological: Placebo (NaCl) — Placebo injection
  Arms: placebo

SUMMARY:
Study drug and dosage form : Umbilical cord-derived mesenchymal stem cells (HB-MSC1)

Dose and route of administration : 60 × 106 cells or 120 x 106 cells to be injected as 30 individual intramuscular injections, once at V0 within 48 hours to 2 weeks maximum after the revascularization procedure.

Comparator, dose and route of administration : Placebo, injected as 30 individual intramuscular injections, once at V2 within 48 hours to 2 weeks maximum after the revascularization procedure.

Study centers : 3 centers in France

Study objectives :

Primary: Evaluation of the feasibility and systemic and local tolerance of an implantation, via intramuscular route, of allogenic HB-MSC1, associated with a revascularization procedure, in patients suffering from critical limb ischemia (CLI).

Secondary: Preliminary evaluation of efficacy and dose effect relationship of the MSC implantation in hemodynamic, anatomical and functional terms.

Exploratory: Constitution of a serum bank of the patients included in the study for inflammation and auto immunity biomarkers analysis

Study design : This will be a multicenter Phase IIa study, consisting in a first, open-label, ascending dose feasibility and safety stage followed by a randomized placebo-controlled feasibility, safety and preliminary efficacy stage.

DETAILED DESCRIPTION:
Demographics, baseline and follow-up characteristics: descriptive statistics. Primary analysis: Descriptive statistics for the rate of patients with high grade AEs (grade 2 and more), related to the cell implantation will be computed in each arm, with its two-sided 95% CIs.

Each dose arm will be compared to the control arm by computing the absolute difference and the relative risk between the active dose arm and the control arm, together with their 95% two-sided CIs.

The p-values for the comparisons of the difference between the observed absolute rate to 0 and of the relative risk to 1 will be computed, but it is not expected that the study will have sufficient power to detect a significant difference on either of the two statistics (absolute difference or relative risk).

Primary efficacy analysis: The primary efficacy criterion (TcPO2) will be compared between each dose group versus the control group to test for a superiority of MSC over control.

The tested hypotheses are:

* Null hypothesis: mean (MSC dose i) ≤ mean (Control)
* Alternative hypothesis: mean (MSC dose i) > mean (Control) A mixed - model for repeated measures will be used to model the evolution of TcPO2 over time. The significance of the time by treatment interaction will be used to test the two hypotheses. Model adjusted means (LS means) and their differences between treatment arms will be computed at each timepoint.

The LS-Means for change from baseline to 180 days will be used as the primary efficacy endpoint.

Other efficacy analyses: the same analysis model (mixed - model for repeated measures) will be used for all the other continuous efficacy endpoints.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is suffering from critical limb ischemia due to atheromatous arteriopathy, and defined as existence of chronic pain at rest or trophic disorders, with a systolic pressure inferior to 50 mm Hg at the ankle or inferior to 30 mm Hg at the toe (respectively 70 and 50 mm Hg in case of trophic disorder), or a transcutaneous measure of oxygen pressure (TcPO2) at the back of the foot in decubitus inferior to 30 mm Hg, and is being subject to a revascularization procedure, associated or not to minimally invasive surgery.

   Inclusion confirmation will be performed after the revascularization procedure, and treatment planned within 48 hours to 2 weeks after the revascularization procedure.
2. The patient (or his/her legal representative(s)) is capable to understand and comply with study requirements and to provide written informed consent prior to any study procedure for participation in the study and transmission of personal "anonymized" data, which signifies an agreement to enter the study and comply with the restrictions and requirements listed in the informed consent form (ICF).
3. Male or female patients aged ≥18 years at the time of signing the ICF.
4. A female patient is eligible to participate if she is of non-childbearing potential, defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or post-menopausal females defined as 12 months of spontaneous amenorrhea. Females on hormone replacement therapy (HRT) will be required to use one of the treatment methods that does not modify hemostasis parameters (eg chlormadinone acetate [Lutéran]) or must discontinue HRT to allow confirmation of post-menopausal status prior to being enrolled in the study.
5. Diabetic patients with an eye fundus examination of less than 3 months excluding proliferative retinopathy
6. Patient with a life expectancy >12 months

Exclusion Criteria:

1. Patients presenting a failure of the revascularization procedure, with technical failure defined as the inability to perform the intended procedure, i.e.

   * in the case where femoropopliteal bypass was intended, inability to perform the bypass for any reason
   * in the case where endovascular procedure was intended:

     * inability to cross the arterial lesion with a guidewire and to catheterize the target vessel
     * inability to cross the arterial lesion with any endovascular treatment device such as balloons or stents
     * residual stenosis > 50%
2. Patient with non atheromatous arteriopathy The patient has, or has a history of, any significant disease or disorder that would increase the risk for the patient if they were enrolled in the study or would affect study procedures or outcomes.
3. The patient is mentally or legally incapacitated.
4. Patient protected by law.
5. Patient who does not benefit from the national health insurance coverage.
6. The patient has been involved in a previous trial with the investigational product.
7. History of cancer excepting basocellular epithelioma during the past 5 years.
8. Patient necessitating chronic hemodialysis or creatinine clearance inferior to 30 mL/min.
9. History of stroke or myocardial infarction of less than 3 months.
10. Hemostasis disorder with contra-indication of intramuscular injections.
11. Patients receiving dual antiplatelet therapy that cannot be temporarily discontinued at least 4 days before and until 6 hours after cell implantation.
12. Patient receiving an antiplatelet therapy with an adenosine diphosphate receptor inhibitor (ADP/P2Y12 inhibitor) that cannot be temporarily discontinued at least 4 days before and until 6 hours after cell implantation.
13. Patient receiving an anticoagulant treatment that cannot be temporarily discontinued until 2 days after the study treatment injection.
14. Patients subject to a below the knee femoro-popliteal bypass procedure or to a femoro-tibial bypass procedure
15. Patients included in another therapeutic trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-09 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment - emergent adverse events | Day 1 to day 360
  The primary safety endpoint will be the occurrence of any high grade AEs (grade 2 and more), either serious or not, assessed as related to the cell implantation by the investigator, reported over the 360 days of the study period.
  AE Intensity Definition :
  Grade 1 : asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated ; Grade 2 : minimal, local or non-invasive intervention indicated; limiting age-appropriate instrumental activities of daily living ; Grade 3 : severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care activities of daily living ; Grade 4 : life-threatening consequences; urgent intervention indicated ; Grade 5 : death related to adverse event

SECONDARY OUTCOMES:
Transcutaneous oxygen pressure | Day 360
  Primary efficacy endpoint: transcutaneous oxygen pressure (TcPO2) mesured in mm Hg

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France